CLINICAL TRIAL: NCT05849116
Title: Effect of High Flow Nasal Cannula Versus Nasal Continuous Positive Airway Pressure on Clinical Outcomes of Preterm Infants With Respiratory Distress Syndrome
Brief Title: Effect of High Flow Nasal Cannula Versus Nasal Continuous Positive Airway Pressure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Noran Hasan Megally, Principal Investigator, Assiut University
Other Study IDs: preterm infants with RDS
Record Dates: First submitted 2023-03-24; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (2):
- High flow nasal cannula: preterms infants who are connected to high flow nasal cannula
- Continuous positive airway pressure: preterms who are connected to continuous positive airway pressure

SUMMARY:
Respiratory distress syndrome (RDS) in preterm babies is caused by a deficiency of lung surfactant. The risk of RDS increases with decreasing gestational age, and is almost inevitable in babies born at less than 28 weeks gestation. Without surfactant the lungs become stiff and the alveoli collapse at end-expiration, and untreated RDS is a major cause of morbidity and mortality in preterm infants

DETAILED DESCRIPTION:
Respiratory distress syndrome (RDS) in preterm babies is caused by a deficiency of lung surfactant. The risk of RDS increases with decreasing gestational age, and is almost inevitable in babies born at less than 28 weeks gestation. Without surfactant the lungs become stiff and the alveoli collapse at end-expiration, and untreated RDS is a major cause of morbidity and mortality in preterm infants Respiratory distress is a common disease in infants, with an incidence rate of 7%, and preterm infants have higher incidences of respiratory distress. Clinical manifestations include apnea, cyanosis, wheezing-like breathing, nasal incontinence, feeding intolerance, shortness of breath or apnea, and inspiratory depression. The most common cause of respiratory distress in preterm infants is neonate respiratory distress syndrome (RDS) Surfactant is a naturally produced surface-active lipoprotein complex mixed with proteins, which reduces the surface tension at the alveolar liquid surface. Surfactant allows alveoli to stay open in expiration and substantially reduces the work of breathing. It also reduces shearing forces on immature alveolar membrane, preventing membrane rupture and protein leak into the alveolar space with resulting lung damage. RDS in preterm babies can be prevented by administration of exogenous animal derived surfactant therapy, and this substantially reduces mortality and respiratory morbidity for this population, including improved survival without bronchopulmonary dysplasia (BPD) at 28 days The use of noninvasive respiratory support, particularly nasal continuous positive airway pressure (nCPAP), has become a common strategy for early respiratory management of preterm infants. In recent years, heated, humidified high-flow nasal cannula (HHHFNC) has increased in popularity in high-resource countries as an alternative form of noninvasive respiratory support for newborn infants. In contrast to nCPAP, for which the rationale is essentially based on the provision of a continuous distending pressure, multiple mechanisms have been suggested to explain HHHFNC functioning, such as washout of the nasopharyngeal dead space, optimal gas conditioning, and provision of a variable distending pressure The HHHFNC approach has been applied in the neonatal intensive care unit (NICU) in a variety of clinical situations: weaning from nCPAP, preventing apnea of prematurity, following extubation, and as primary therapy for respiratory distress syndrome (RDS). Compared with nCPAP, HHHFNC offers ease of use, reduced risk of nasal injuries, better infant tolerance with improved feeding, and bonding HFNC works by providing inhaled gases at flows higher than the inspiratory demand flow. This leads to wash out of upper airways, reduces physiological dead space, and decreases nasopharyngeal airway resistance. It also provides variable positive end expiratory pressure and decreases work of breathing. But, as delivering HFNC requires a loose-fitting nasal prong, the pressure delivery is not reliable. The three important components of HFNC include a flow generator, an air-oxygen blender, and a heater-humidifier. HFNC has gained popularity because of the ease of use, lesser nasal trauma, and more comfort to the neonate Nasal CPAP is a method of delivering nasopharyngeal pressure to a spontaneously breathing neonate, where pressure is maintained throughout the respiratory cycle (both inspiration and expiration). Nasal CPAP works by decreasing airway resistance, increasing functional residual capacity, stabilizing chest wall, and splinting the airway (upper and lower). The preventive use of nasal CPAP (nCPAP) in preterm infants declines the need for mechanical ventilation and ultimately, reduces the rate of pneumothorax and mortality, especially accompanied with surfactant administration Invasive mechanical ventilation is widely used in neonatal intensive care units (NICUs). However, long-term invasive mechanical ventilation can lead to ventilator-related lung injuries, including pressure injuries, volume injuries, and ventilator pneumonia. In later stages, it may even lead to severe infection and bronchopulmonary dysplasia (BPD) The objective of the study was to evaluate the effect of high flow nasal cannula versus CPAP on the clinical outcomes of preterm infants with respiratory distress syndrome

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants ≥30 weeks
* Preterm infants with birth weight >1000 gm
* Preterm infants diagnosed with respiratory distress syndrome.

Exclusion Criteria:

1. Full term infants (>37 weeks)
2. Preterm infants (<30 weeks & less than 1000 gm)
3. Neonates with respiratory distress other than respiratory distress syndrome.
4. Neonates with neonatal sepsis.
5. Neonates with congenital anomalies including congenital heart diseases.
6. Neonates who need invasive MV immediately after birth.

Ages: 30 Weeks to 37 Weeks | Sex: All
Age Groups: Child
Study Population: 100 preterm infants between 30 weeks and 37 weeks
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
The rate of invasive mechanical ventilation at the first 72 hours of life. | first 72 hours of life
  Regarding the following aspect:
  The effect of high flow nasal cannula versus CPAP on the clinical outcomes of preterm infants with respiratory distress syndrome regarding the need for invasive mechanical ventilation at the first 72 hours of life.
Time for weaning off from oxygen. | Baseline
  Regarding the following aspect:
  The effect of high flow nasal cannula versus CPAP on the clinical outcomes of preterm infants with respiratory distress syndrome regarding the time for weaning off from oxygen.
Duration of hospital stay. | Baseline
  Regarding the following aspect:
  The effect of high flow nasal cannula versus CPAP on the clinical outcomes of preterm infants with respiratory distress syndrome regarding the duration of hospital stay.
Rate of morbidity and mortality. | Baseline
  Regarding the following aspect:
  The effect of high flow nasal cannula versus CPAP on the clinical outcomes of preterm infants with respiratory distress syndrome regarding the effect on morbidity and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Gafar Ibrahim, Prof, Principal Investigator — Assiut University; Safwat Moahmed, Assist prof, Principal Investigator — Assiut University